CLINICAL TRIAL: NCT06989320
Title: Endogenous Oxalate Synthesis in Idiopathic Calcium Oxalate Kidney Stone Formers
Brief Title: Endogenous Oxalate Synthesis in Idiopathic Calcium Oxalate Kidney Stone Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of Texas, Southwestern Medical Center at Dallas (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Sonia Fargue, Associate professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB300014279-OSS; R01DK137784 (NIH)
Record Dates: First submitted 2025-05-09; First posted 2025-05-25 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Kidney Stones; Kidney Calculi; Urolithiasis; Urolithiasis, Calcium Oxalate; Nephrolithiasis; Nephrolithiasis, Calcium Oxalate; Oxalate Urolithiasis; Healthy; Healthy Volunteer
Keywords: oxalate synthesis
MeSH Terms: conditions — Kidney Calculi; Urolithiasis; Nephrolithiasis, Calcium Oxalate; Nephrolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Idiopathic Calcium Oxalate Kidney Stone Patients (Experimental): Low oxalate fixed diets. oral glycolate and ascorbic acid administration
  Interventions: Dietary Supplement: Low-oxalate diet and glycolate dosing; Dietary Supplement: Oral glycolate dosing; Dietary Supplement: Oral 13C- ascorbic acid dosing
- Healthy non-kidney stone forming individuals (Active Comparator): Low oxalate fixed diets. oral glycolate and ascorbic acid administration
  Interventions: Dietary Supplement: Low-oxalate diet and glycolate dosing; Dietary Supplement: Oral glycolate dosing; Dietary Supplement: Oral 13C- ascorbic acid dosing

INTERVENTIONS:
Dietary Supplement: Low-oxalate diet and glycolate dosing — Low-oxalate diet 4 days of fixed eucaloric diet with low oxalate (<60 mg/day), normal calcium content (600-1000 mg/day)
Dietary Supplement: Oral glycolate dosing — Oral 13C-glycolate dosing (0.5 mg/kg)
Dietary Supplement: Oral 13C- ascorbic acid dosing — Oral 13C- ascorbic acid dosing (0.75 mg/kg)

SUMMARY:
The goal of this clinical trial study is to test if patients with idiopathic calcium oxalate kidney stones have an increased production of oxalate by the body, which would lead to increased urinary excretion of oxalate.

The study will recruit adult patients with a history of calcium oxalate kidney stones and healthy volunteers without kidney stones.

Participants will

ingest fixed diets containing low amounts of oxalate for 5 days ingest a soluble form of glycolate and vitamin C collect urine, blood, stool during the dietary and oral dosing portions of the study and also collect breath sample during the oral glycolate test

DETAILED DESCRIPTION:
In this study the investigators propose to measure the production of oxalate by the body (endogenous oxalate synthesis), after equilibration on a low oxalate diet (<60 mg oxalate/day, 600-800 mg calcium/day) and estimate the importance of vitamin C and glycolate metabolism to oxalate production in both Calcium Oxalate Kidney Stone patients and matched controls by oral dosings of those two substances.

Phase 1. Screening and low-oxalate diet 24-hr urinary excretions. Between the University of Alabama at Birmingham (UAB) and the University of Texas Southwestern Medical Center (UTSW), the study will enroll 40 subjects with idiopathic Calcium Oxalate Kidney Stone (20 Males/20 Females) and 40 non-kidney stone forming controls (20 Males/20 Females). Participants in the two groups will be matched for age (within 10 yrs) and gender. Screening will include blood complete metabolic profile and two 24-hour urine specimens collected at home on self-choice diets and anthropometric measurements.

Participants will then ingest the controlled low-oxalate (<60 mg/day) diet for 5 consecutive days and collect two 24-hour urines after 2 days of dietary equilibration.

Phase 2. Oxalate production and 13C-glycolate dosing tests. On Day 5, participants will arrive after an overnight fast in the research unit to undergo the oral 13C-glycolate dosing test. After a 1-hour baseline urine collection, they will ingest an oral load containing 0.5 mg/kg body weight of 13C-glycolate, dissolved in bottled water. For the next 7 hours, blood and urine will be collected hourly, and breath as more time points. They will remain on the fixed diet for 24 hours with a meal 7 hours post-load, and dinner at home 12 hours post-load. They will collect the remainder of their 24-hour urine at home.

Phase 3. Oxalate production and 13C-ascorbic acid dosing tests. After 1 day of equilibration on the same low-oxalate diet, participants will arrive after an overnight fast in the research unit to provid eone blood and one urine sample and then ingest an oral dose of 13C-ascorbic acid (0.75 mg/kg), return home and continue to ingest the low-oxalate diet. The next morning, participants will arrive after an overnight fast in the research unit. For the next 7 hours, blood and urine will be collected hourly. They will remain on the fixed diet for 24 hours with a meal at the end of the visit.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 yrs
* Body Mass Index > 18.5 kg/m2
* Normal fasting serum electrolytes on comprehensive metabolic profile
* Willing to ingest fixed diets
* Willing to stop supplements (vitamins including vitamin C, calcium (citrate or carbonate) and other minerals, herbal supplements, nutritional aids, probiotics) for 2 weeks before start and during study.
* For stone formers: first time or recurrent Calcium Oxalate stone former. Composition of most recent stone ≥ 50% calcium oxalate if available, uric acid component <20%

Exclusion Criteria:

* Chronic Kidney Disease stage 4-5
* Primary hyperoxaluria, Enteric (secondary) hyperoxaluria
* Liver, bowel, endocrine or renal diseases (other than idiopathic Calcium Oxalate kidney stones) or any other condition that may influence the absorption, transport or urinary excretion of ions, which will compromise the interpretation of results, including: Cystic fibrosis, Celiac disease, Cystinuria, Uric acid stone former, Nephrotic syndrome, Sarcoidosis, Renal tubular acidosis, Primary hyperparathyroidism, Neurogenic bladder, Urinary diversion, Chronic diarrhea, Bariatric surgery, Inflammatory bowel disease
* Pregnancy or breast-feeding
* Incompatible dietary requirements with the study, food allergies or intolerance to any of the foods in study menus
* Active malignancy or treatment for malignancy within 12 months prior to screening
* Utilization of immunosuppressive medication
* Uncontrolled hypertension or diabetes
* Diabetes type 1

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Estimated endogenous oxalate synthesis (oxalate mg/day) | 1 day
  Basal rate of endogenous oxalate synthesis estimated by repeat fasted hourly urine collections (mg/day)

SECONDARY OUTCOMES:
24-hour urinary oxalate excretion on low oxalate diet | 2 days
  mean 24-hour urinary oxalate excretion on the low oxalate diet (mg/day)
contribution of ascorbic acid breakdown to urinary oxalate excretion | 2 days
  contribution of ascorbic acid breakdown to oxalate synthesis (%)

OTHER OUTCOMES:
Contribution of glycolate metabolism to urinary oxalate | 1 day
  Proportion of 13C-glycolate orally dosed that is metabolized to urinary 13C-oxalate in the fasted stated (%)

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Fargue, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - United States, Alabama University of Alabama at Birmingham, Birmingham, Alabama
  - University of Texas South Western Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No